CLINICAL TRIAL: NCT00193271
Title: Adjuvant Chemotherapy (Docetaxel and Estramustine Phosphate) for High Risk Localized Prostate Cancer
Brief Title: Adjuvant Docetaxel and Estramustine Phosphate for High Risk Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: SCRI Oncology Research Consortium, SCRI
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 19; IIT16165
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Estramustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Docetaxel
Drug: Estramustine

SUMMARY:
This trial will evaluate the feasibility, toxicity, and efficacy of docetaxel/estramustine, as in the adjuvant therapy of patients with high-risk prostate cancer after definitive local therapy.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will receive:

Docetaxel + Estramustine

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Clinically or surgically staged localized disease, stage I-III.
* Prior surgical resection or radiation therapy with curative intent
* No clinical evidence of residual disease
* Gleason's combined score > 7.
* Age > 18 years.
* No prior chemotherapy for prostate cancer.
* No previous androgen deprivation therapy for prostate cancer
* Able to perform activities of daily living with minimal assistance
* Adequate bone marrow, liver and kidney function
* Voluntarily provide written informed consent.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* History of prior malignancy in the past five years
* History of significant heart disease within the previous 6 months
* Cerebral vascular accident (CVA) or stroke within the previous 6 months.
* Moderate or severe peripheral neuropathy
* Previous therapy with other injectable radioisotopes.

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Response Rate

SECONDARY OUTCOMES:
Rate of recurrence
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Anthony A. Meluch, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States